CLINICAL TRIAL: NCT04133870
Title: Exploratory Study of the Molecular Profile of Thyroid Cancer
Brief Title: Identification of Molecular Biomarkers for Thyroid Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4343
Record Dates: First submitted 2017-01-26; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2018-11

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour tissue for NGS panel testing. The tissue will be routinely processed formalin fixed paraffin embedded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a two part study; part A proposes to collect plasma samples to examine how ctDNA (circulating thyroid DNA) markers correlate with detection of recurrent disease, response to therapy, clinical outcome and pathological data. Part B aims to use tissue obtained from biopsies of primary or recurrent disease to establish cell lines and tumour explants to further investigate the biology of thyroid cancer in the preclinical setting

DETAILED DESCRIPTION:
To collect blood and tumour tissue for Part A: molecular profiling, including extraction of DNA for sequencing, RNA for expression levels and to identify expressed fusion genes, and proteins for proteomic studies and Part B: for establishment of cell lines and patient derived xenograft (PDX) models of thyroid cancer.

1. To correlate BRAF V600E, RAS, RET/PTC, RET, PAX8/PPARϒ, βcatenin, p53, PTEN and PI3K mutations in ctDNA with Formalin Fixed Paraffin Embedded tumour tissue (FFPE) mutational analysis.
2. To correlate the quantity of ctDNA fragments 3 monthly in patients with advanced disease on routine follow up with conventional tumour markers (Tg, calcitonin, CEA).
3. To correlate the quantity of ctDNA fragments 3 monthly once relapse suspected by conventional methods (Tg, Calcitonin, CEA, radiological)
4. To correlate the quantity of ctDNA fragments with response (RECIST, Tg, Calcitonin and CEA) to targeted therapies
5. To assess prognostic significance of ctDNA levels in metastatic/advanced thyroid cancer
6. To isolate live tumor cells for studies of novel treatment strategies (combinatorial treatments), therapy resistance and thyroid cancer biology
7. Retrieval and analysis of archival primary tissue blocks for comparison with metastatic tumour sites
8. To collect blood for analysis of noninvasive tests of tumour phenotype

ELIGIBILITY:
Inclusion Criteria:

* T3-4, N0-1b, M0-M1 thyroid cancer (papillary, follicular, poorly differentiated, anaplastic and medullary thyroid carcinoma).
* Patient able to provide informed consent
* Patient attending the Royal Marsden Hospital for inpatient or outpatient review
* Sufficient tissue sample available to perform analysis (archived or fresh)
* Adults >16 years old

Exclusion Criteria:

* Patients unable to provide informed consent
* Thyroid lymphoma
* Metastases to the thyroid
* No histological confirmed diagnosis
* Only cytology available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a biological study to obtain tissue and blood samples from patients with advanced thyroid cancer
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 3 Years (at the end of study)
  Part A: blood and tumour tissue will be measured to determine molecular profiling.
Primary Objective | 3 years (at end of study)
  Part B: blood and tumour tissue will be assessed to establish cell lines and to determine patient derived xenograft (PDX) models of thyroid cancer

CONTACTS AND LOCATIONS:
Overall Officials: Kate Newbold, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, London, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided